CLINICAL TRIAL: NCT02442531
Title: A Phase I Open-Label, Safety, Pharmacokinetic and Preliminary Efficacy Study of CriPec® Docetaxel in Patients With Solid Tumours
Brief Title: A Study of CriPec® Docetaxel Given to Patients With Solid Tumours
Acronym: NAPOLY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cristal Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-CL01
Record Dates: First submitted 2015-05-01; First posted 2015-05-13 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-07

CONDITIONS: Cancer; Metastatic Cancer; Solid Tumors
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CriPec® docetaxel (Experimental): Docetaxel containing nanoparticle
  Interventions: Drug: CriPec® docetaxel

INTERVENTIONS:
Drug: CriPec® docetaxel — -3 weekly IV dose. Dose escalation; start dose 15 mg/m2. Number of cycles: 6 or until progression or unacceptable toxicity develops
  Other Names: Docetaxel containing nanoparticles

SUMMARY:
The goal of this Phase1 clinical research study is to find the highest safe dose of CriPec® docetaxel that can be given in the treatment of patients with solid tumours.

DETAILED DESCRIPTION:
The study is designed to explore the safety, tolerability, pharmacokinetics and pharmacodynamics of CriPec® docetaxel and to identify the Maximum Tolerated Dose (MTD).

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
3. Estimated life expectancy of at least 12 weeks
4. Ability and willingness to give written informed consent and to comply with the requirements of the study

   For Part 1:
5. Patients with pathologically confirmed diagnosis of advanced, recurrent and progressive solid tumours that are refractory to standard therapy or for whom no standard therapy exists and with measurable or evaluable disease according to RECIST 1.1.

   For Part 2:
6. Patients with pathologically confirmed diagnosis of advanced, recurrent and progressive cancer with measurable disease according to RECIST 1.1 of a histological type that are refractory to standard therapy or for whom no standard therapy exists and where treatment with a taxane is an appropriate treatment option.

Exclusion Criteria:

1. Less than 4 weeks since the last treatment of chemotherapy, biological therapy, immunotherapy or systemic radiotherapy (except palliative radiation delivered to <20% of bone marrow), and less than 6 weeks for nitrosoureas and mitomycin C prior to Cycle 1 Day 1.
2. Current or recent (within 4 weeks prior to Cycle 1 Day 1) treatment with another Investigational Product or participation in another investigational interventional study.
3. Symptomatic brain metastases.
4. Toxicities incurred as a result of previous anticancer therapy (radiation therapy, chemotherapy, or surgery) that have not resolved to ≤ grade 2 (as defined by CTCAE version 4.03).
5. Inadequate bone marrow function at screening as evidenced by any of the following:

   * Absolute Neutrophil Count (ANC) < 1.5 x 109/L.
   * Platelet count < 100 x 109/L.
   * Haemoglobin < 6.0 mmol/L (< 9.6 g/dL). The patient should not have received a transfusion or growth factors for these abnormalities in the 7 days prior to Cycle 1 Day 1.
6. Serum (total) bilirubin > 1.5 x the Upper Limit of Normal (ULN) for the institution if no liver metastases (> 2 x ULN in patients with liver metastases).
7. AST or ALT > 2.5 x ULN if no liver metastases (> 5x ULN in patients with liver metastases).
8. Alkaline phosphatase levels > 2.5 x ULN if no liver metastases (> 5 x ULN in patients with liver metastases, or > 10 x ULN in patients with bone metastases).
9. Increased plasma prothrombin time or International Normalized Ratio (INR), consequence of reduced hepatic production of Vitamin K.
10. Hepatitis B surface antigen or hepatitis C positivity with abnormal liver function tests.
11. Medical history of:

    * Nonalcoholic steatohepatitis (NASH).
    * History of human immunodeficiency virus (HIV) antibody positive or use of antiretroviral therapy.
    * Alcoholic and autoimmune hepatitis.
    * Ischemic hepatitis, Cardiovascular dysfunction or impaired liver oxygenation, including hypotension or right heart failure.
12. Serum creatinine > 1.5 x ULN.
13. Estimated Glomerular Filtration Rate of < 50 mL/min/1.73m2 calculated by Modification of Diet in Renal Disease (MDRD) formula or creatinine clearance of < 50 mL/min calculated by Cockcroft-Gault.
14. Stroke within 6 months prior to Cycle 1 Day 1.
15. Transient Ischemic Attack (TIA) within 6 months prior to Cycle 1 Day 1.
16. Myocardial infarction within 6 months prior to Cycle 1 Day 1.
17. Unstable angina.
18. New York Heart Association (NYHA) Grade II or greater Congestive Heart Failure at screening.
19. Serious cardiac arrhythmia requiring medication.
20. Patients who are pregnant or breastfeeding.
21. Absence of effective means of contraception in female patients of childbearing potential (defined as <2 years after last menstruation and not surgically sterile) or in male patients who are not surgically sterile and who have female partners of childbearing potential.
22. Major surgical procedure (including open biopsy and excluding central line intravenous catheter) within 28 days prior to the first study treatment, or anticipation of the need for major surgery during the course of the study treatment.
23. Grade ≥2 motor or sensory neuropathy symptoms (as defined by CTCAE version 4.03).
24. Known hypersensitivity to any of the Investigational Product's excipients or taxanes.
25. History of drug or alcohol abuse in the opinion of the investigator within 3 years before screening.
26. Evidence of any other medical conditions (such as psychiatric illness, infectious diseases, physical examination or laboratory findings) that may interfere with the planned treatment, affect patient compliance or place the patient at high risk for treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Part 1: Incidence of grade 3 or 4 adverse events (AEs) as a measure of safety and tolerability. | 9 months
  Part 1: Incidence of grade 3 or 4 adverse events (AEs) will be determined after escalating doses of CriPec® docetaxel once every three weeks.
Part 1: Incidence of clinical laboratory abnormalities as a measure of safety and tolerability. | 9 months
  Part 1: Incidence of laboratory abnormalities will be determined after escalating doses of CriPec® docetaxel once every three weeks.
Part 1: Incidence of electrocardiogram (ECG) abnormalities as a measure of safety and tolerability. | 9 months
  Part 1: Incidence of electrocardiogram (ECG) abnormalities will be determined after escalating doses of CriPec® docetaxel once every three weeks.
Part 2: Incidence of grade 3 or 4 adverse events (AEs) at the Maximum Tolerated Dose (MTD) of CriPec® docetaxel as defined in Part 1. | 9 months
  Part 2: Incidence of grade 3 or 4 adverse events (AEs) at the Maximum Tolerated Dose will be determined after CriPec® docetaxel dosing once every three weeks.
Part 2: Incidence of clinical laboratory abnormalities at the Maximum Tolerated Dose (MTD) of CriPec® docetaxel as defined in Part 1 | 9 months
  Part 2: Incidence of clinical laboratory abnormalities at the Maximum Tolerated Dose will be determined after CriPec® docetaxel dosing once every three weeks.
Part 2: Incidence of electrocardiogram (ECG) abnormalities at the Maximum Tolerated Dose (MTD) of CriPec® docetaxel as defined in Part 1 | 9 months
  Part 2: Incidence of electrocardiogram (ECG) abnormalities at the Maximum Tolerated Dose will be determined after CriPec® docetaxel dosing once every three weeks.
Part 1 and 2: Pharmacokinetic profile of CriPec® docetaxel following IV infusion | First two cycles of CriPec® docetaxel (each cycle is 3 weeks)
  Pharmacokinetic parameters such as time to peak concentration (Tmax), peak concentration (Cmax), volume of distribution (Vd), half life (t1/2), total body clearance (CL) and area under the concentration-time curve (AUC) will be determined using plasma concentration data.

SECONDARY OUTCOMES:
Early signs of anti-tumor efficacy (overall response rate [ORR]) of CriPec® docetaxel | 18 months in total for part 1 and 2
Early signs of anti-tumor efficacy (duration of response) of CriPec® docetaxel | 18 months in total for part 1 and 2

CONTACTS AND LOCATIONS:
Locations (4):
- University Hospital Leuven, Leuven, Belgium
- Netherlands (3):
  - VUMC Amsterdam, Amsterdam
  - UMC Groningen, Groningen
  - Erasmus Medical Center, Rotterdam